CLINICAL TRIAL: NCT06138093
Title: Consequence of Open Versus Closed Tracheostomy Immediately After Decannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 74553
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2023-11

CONDITIONS: Tracheostomy
Keywords: tracheostomy; respiratory insufficiency; respiratory function tests; mechanical ventilators; rehabilitation; critical care
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sealed / closed tracheostomy (Experimental): Sealing of the tracheostomy wound using a sealing device.
  Interventions: Device: Sealing device; Device: No device

INTERVENTIONS:
Device: Sealing device — Intratracheal tracheostomy sealing
Device: No device — Open tracheostomy wound

SUMMARY:
Tracheostomy is performed for prolonged mechanical ventilation. Ineffective bandaging following decannulation leaves the tracheostomy wound unsealed, reducing pulmonary function, coughing ability, and voice quality, ultimately leading to decannulation failure. Recently, a new concept enabling intratracheal sealing of the tracheotomy was introduced, potentially solving the issues of air leakage and tracheal wound infection. This study aims to investigate the feasibility of intratracheal tracheostomy sealing in relation to an immediate normalization of physiological airway flow and an improved voice quality.

DETAILED DESCRIPTION:
See protocol document.

ELIGIBILITY:
Inclusion Criteria:

* Tracheostomy for minimum 7 days
* Age > 18 years
* Capped uncuffed tube size 7 or 8 for at least 24 hours

Exclusion Criteria:

* Cognitive dysfunction (patients who are not able to cooperate with investigation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | Day 2: At time of decannulation, i.e. directly after inclusion and randomization to sealing or not as first intervention
  Lung function / air flow evaluated by spirometry
Voice quality | Day 2: At time of decannulation, i.e. directly after inclusion and randomization to sealing or not as first intervention
  Evaluated by Equal-Appearing Interval Scale ranging from 1 to 5, where 5 represents a normal voice quality and 1 represents a severely impaired voice
Peak expiratory flow (PEF) | Day 2: At time of decannulation, i.e. directly after inclusion and randomization to sealing or not as first intervention
  Lung function / air flow evaluated by spirometry
Forced vital capacity (FVC) | Day 2: At time of decannulation, i.e. directly after inclusion and randomization to sealing or not as first intervention
  Lung function / air flow evaluated by spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus E Kraghede, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care, Aarhus University Hospital; J. Michael Hasenkam, MD, DMSc, Study Chair — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital
Locations (1):
- Department of Anaesthesiology and Intensive Care, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraghede RE, Christiansen KJ, Kaspersen AE, Pedersen M, Petersen JJ, Hasenkam JM, Devantier L. Novel Method for Sealing Tracheostomies Immediately after Decannulation-An Acute Clinical Feasibility Study. Biomedicines. 2024 Apr 12;12(4):852. doi: 10.3390/biomedicines12040852. PMID 38672206

DOCUMENTS (1):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT06138093/Prot_000.pdf